CLINICAL TRIAL: NCT04015778
Title: A Two-arm (Phase 2) Exploratory Study of Nivolumab Monotherapy or in Combination With Nab-paclitaxel and Carboplatin in Early Stage NSCLC in China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG 1804
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Carboplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab Mono (Experimental): In arm A, 24 participants will be enrolled into this arm according to PD-L1 expressing level (≥50%).Arm A consists of 3 cycles of neoadjuvant nivolumab (240mg every 2 weeks), and adjuvant nivolumab (240mg IV, over 30 min, every 2 weeks) up to 12 months
  Interventions: Biological: Nivolumab
- Nivolumab Plus Chemo (Experimental): In arm B, up to 12 participants will be enrolled into each subgroup according to PD-L1 expressing level (<1% and 1%-49%).arm B consists of 3 cycles of neoadjuvant nivolumab (360mg every 3 weeks) with nab-paclitaxel and carboplatin(nab-paclitaxel 135 mg/m2, d1, 8 and carboplatin AUC 5, d1 every three weeks ), and adjuvant nivolumab (240mg IV, over 30 min, every 2 weeks) up to 12 months
  Interventions: Biological: Nivolumab; Drug: carboplatin; Drug: nab-paclitaxel

INTERVENTIONS:
Biological: Nivolumab — 240mg Q2W or 360mg Q3W
Drug: carboplatin — AUC 5, d1 every three weeks
  Arms: Nivolumab Plus Chemo
Drug: nab-paclitaxel — 135 mg/m2, d1, 8
  Arms: Nivolumab Plus Chemo

SUMMARY:
Nivolumab (BMS-936558) is a fully human, IgG4 (kappa) isotype mAb that binds PD-1 on activated immune cells and disrupts engagement of the receptor with its ligands PD-L1 (B7 H1/CD274) and PD-L2 (B7-DC/CD273), thereby abrogating inhibitory signals and augmenting the host antitumor response. In early clinical trials, nivolumab has demonstrated activity in several tumor types, including melanoma, renal cell carcinoma (RCC), and non-small cell lung cancer (NSCLC).

Nivolumab is in clinical development for the treatment of patients with NSCLC, RCC, melanoma, squamous cell carcinoma of the head and neck (SCCHN) and other tumors (eg, glioblastoma multiforme, mesothelioma, small cell lung cancer, gastric).

Nivolumab is approved in the United States (US), European Union, and other countries for the treatment of patients with unresectable or metastatic melanoma, advanced NSCLC with progression on or after platinum-based chemotherapy, advanced RCC whose disease progressed on an antiangiogenic therapy, classical Hodgkin lymphoma that has relapsed or progressed after autologous hematopoietic stem cell transplantation and post-transplantation brentuximab vedotin treatment, and recurrent or metastatic squamous cell carcinoma of the head and neck with disease progression on or after a platinum-based therapy.

The proposed study will evaluate the efficacy and safety of preoperative administration of Nivolumab or Nivolumab combined with nab-paclitaxel and carboplatin in neoadjuvant setting and administration of Nivolumab in adjuvant setting in patients with high-risk resectable NSCLC, and will facilitate a comprehensive exploratory characterization of the tumor immune microenvironment and circulating immune cells in these patients. Data obtained in this study will provide valuable information for planning further prospective clinical trials of anti-PD-1 and other immunotherapies in NSCLC, both in the peri-operative and advanced disease setting. Ultimately, it is highly desirable to discover prospective biomarkers of response and toxicity to allow patients with NSCLC who are most likely to derive benefit to receive anti-PD-1 treatment, and conversely to minimize the risk of toxicity and ineffective treatment for patients who are unlikely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Early stage IB-IIIA, operable non-small cell lung cancer, confirmed in tissue
* Lung function capacity capable of tolerating the proposed lung surgery
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Available tissue of primary lung tumor

Exclusion Criteria:

* Presence of locally advanced, inoperable or metastatic disease
* Participants with active, known or suspected autoimmune disease
* Prior treatment with any drug that targets T cell co-stimulations pathways (such as checkpoint inhibitors)

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
MPR rate | The patients considered to be technically resectable will undergo resection，an expected average of 13 weeks
  MPR rate, defined as number participants with <10% residual tumor in lung and lymph nodes, divided by the number of treated participants for each arm Viable tumors in situ carcinoma should not be included in MPR calculation.

SECONDARY OUTCOMES:
MPR rate in 2 subgroups patients (PD-L1 <1%, and 1-49%) in Arm B | The patients considered to be technically resectable will undergo resection，an expected average of 13 weeks
Proportion of resection without delay | The patients considered to be technically resectable will undergo resection，an expected average of 13 weeks
Number of Participants with Adverse Events | During the neoadjuvant period and 100 days post adjuvant period
  Safety and tolerability will be measured by incidence of AE, SAE, immune related AEs, deaths, and laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu SY, Dong S, Yang XN, Liao RQ, Jiang BY, Wang Q, Ben XS, Qiao GB, Lin JT, Yan HH, Yan LX, Nie Q, Tu HY, Wang BC, Yang JJ, Zhou Q, Li HR, Liu K, Wu W, Liu SM, Zhong WZ, Wu YL. Neoadjuvant nivolumab with or without platinum-doublet chemotherapy based on PD-L1 expression in resectable NSCLC (CTONG1804): a multicenter open-label phase II study. Signal Transduct Target Ther. 2023 Dec 6;8(1):442. doi: 10.1038/s41392-023-01700-4. PMID 38057314